CLINICAL TRIAL: NCT04750707
Title: Hydroxyurea Therapy for Neurological and Cognitive Protection in Pediatric Sickle Cell Anemia in Uganda: A Single Arm Open Label Trial, "BRAIN SAFE II"
Brief Title: Hydroxyurea Therapy for Neurological and Cognitive Protection in Pediatric Sickle Cell Anemia in Uganda ( BRAINSAFE-II )
Acronym: BRAINSAFEII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Global Health Uganda LTD (Other)
Collaborators: Columbia University (Other); University of Pittsburgh (Other); Emory University (Other); Mulago Hospital, Uganda (Other); Makerere University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REC REF 2019-147; R01HD096559 (NIH)
Record Dates: First submitted 2021-01-25; First posted 2021-02-11 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Sickle Cell Anemia in Children
MeSH Terms: interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm (Other): Single arm, open label of hydroxyurea starting at 20mg/kg and increased to 30mg/kg depending on clinical need and according to standard guidelines
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea — The study intervention will be daily oral Hydroxyurea given in single doses starting at approximately 20mg/kg/day and escalated to a maximum 30mg/kg/day depending on clinical need and according to standard guidelines.
  Other Names: Siklos

SUMMARY:
Worldwide, an estimated 200,000 babies are born with Sickle Cell Anemia (SCA) annually. Affected children suffer chronic ill health with some having frequent hospitalization. The patients are also at a high risk of brain injury arising from small and large cerebral blood vessel damage in SCA, also called sickle cell vasculopathy (SCV). SCV is associated with the high risk of stroke. Such injury may manifest with neurological and cognitive impairment. An abnormal blood flow to the brain, as measured by a Doppler Ultrasound scan is a known risk factor for stroke.

The hypothesis is that hydroxyurea therapy will prevent, stabilize or improve SCV and its effects.

The study is an open label, single arm clinical trial to test the impact of hydroxyurea treatment in 270 children with SCA starting at ages 3-9 years.

Following baseline assessments, all participants will begin hydroxyurea therapy starting at about 20mg/kg/day. Changes in the frequency and severity of each test (neurological and cognitive tests and cerebral blood flow velocity) will be compared with their baseline tests (prior to hydroxyurea) by repeating these tests at 18 and 36 months. In a randomly selected subset of 90 participants, an evaluation of the impact of hydroxyurea on structural brain vascular injury using magnetic resonance brain imaging (MRI) and magnetic vessel imaging ,also called angiography (MRA) at baseline and at 36 months. Lastly, an assessment of changes to biomarkers of anemia, inflammation and malnutrition from before and during hydroxyurea therapy and determine their relationship to the outcomes. The proposed intervention with hydroxyurea is the first Africa-based trial to broadly prevent or ameliorate manifestations of SCV.

DETAILED DESCRIPTION:
Annually, an estimated 200,000 babies are born with Sickle Cell Anemia (SCA) worldwide. Affected children often suffer repeated acute illnesses and chronic ill health from vascular occlusive phenomenon. In particular, they are at a high risk of stroke due to the development of sickle cell cerebral vascular (SCV) injury. SCV can also cause neurocognitive impairment. Stroke risk may be predicted by abnormal cerebral arterial flow detected by transcutaneous Doppler ultrasound (TCD).

The specific aims are:

Aim 1: Determine the impact of hydroxyurea therapy on the frequency and severity of SCV in a cohort of children treated for three years, as measured by 3 distinct outcomes: abnormal TCD, neurocognitive impairment and primary stroke, compared with baseline.

Aim 2: Evaluate the impact of hydroxyurea on structural SCV using MRI and MRA in a randomly selected subset of this cohort.

Aim 3: Assess changes to anemia, malnutrition status, C-reactive protein and other inflammatory markers during hydroxyurea therapy, over time, compared with baseline levels.

Design: This will an open label, single arm trial of hydroxyurea to test the three year impact of hydroxyurea treatment in children with SCA on each of three clinically important outcomes: abnormal cerebral arterial flow, neurocognitive impairment and primary stroke.

In aim 1, there will be enrollment of a new longitudinal cohort of 270 children ages 3-9 years selected randomly from among eligible patients attending Mulago hospital SCA clinic (MHSCC) roster, without evidence of prior stroke by examination. The hypothesis is that hydroxyurea therapy will prevent, stabilize or improve Sickle Cell Vasculopathy(SCV) and its effects. Eligible subjects will be evaluated by TCD, stroke-focused neurological examination and neurocognitive testing at baseline. Following initial assessments, study subjects will begin standardized hydroxyurea therapy. Overtime, changes in the frequency and severity of each distinct measure of SCV with baseline by repeating these three tests at 18 and 36 months and against the age specific prevalence of SCV in children who did not receive any intervention in the earlier BRAIN SAFE I observational study (our historical cohort).

In Aim 2, a subset of the study subjects, a randomly selected subset of 90 subjects, will undergo brain imaging at baseline and at 36 months to assess structural findings over time. The hypothesis is that prospective brain imaging by MRI and MRA provides critical structural definitions [1,2] of SCV changes or stabilization over three years compared to baseline, while on hydroxyurea. Results of brain imaging and biomarkers will be correlated with these outcomes over time.

In aim 3, there will be prospective examination for risk factors of SCV overtime. Biomarkers for risk of SCV may include severe anemia, the inflammatory marker C- reactive protein (CRP) and malnutrition status. The hypothesis is that a higher burden of anemia, inflammation and malnutrition predispose African children with SCA to greater burden of SCV than in the West. Changes in the values of these biomarkers will be assessed over time while on hydroxyurea

Site: Participants will be recruited from Mulago hospital Sickle Cell Anemia Clinic in Kampala, Uganda.

Follow up: Participants will be on study medication and follow-up for 36 months.

Data Analysis: The investigators will estimate the effects of hydroxyurea for each distinct endpoint, (stroke, abnormal TCD or impaired cognition) by comparing against the age specific prevalence in children who did not receive any intervention in the earlier BRAIN SAFE I study. To assess the risk of stabilization or reduction in SCV, time to event analyses using Cox proportional hazards modelling will be used after Kaplan Meier curves are generated. Multilevel regression models will be used to asses within and between subject changes over time for continuous measures of TCD velocity and cognitive z-scores.

ELIGIBILITY:
Inclusion Criteria:

1. Documented laboratory diagnosis of HbSS or HbS-B 0 thalassemia (both types are treated equally in SCA studies)
2. Ages 3 through 9 years (inclusive) at enrolment
3. To ensure clinic follow-up, child has attended Mulago Hospital Sickle Cell Anaemia (SCA)clinic 2 times in the prior 4 years, or at least once in the past 2 years if younger than < 4 years
4. No history of hydroxyurea use for longer than 6 months
5. Parent/legal guardian has provided a written consent (and if child is ≥8 years of age, has provided assent)

Exclusion Criteria:

1. History of neurological abnormality known before age 4 months (to avoid those with non SCA brain injury)
2. Child is currently enrolled in another clinical intervention trial
3. Prior stroke as detected by standard Pediatric NIH Stroke Scale (PedNIHSS) examination

   Temporary exclusion criteria
4. Pre-existing hematological toxicity

   1. Hemoglobin <4.0 gm/dL
   2. Hemoglobin <6.0 gm/dL with Absolute Reticulocyte Count <100 x 10 9/L
   3. Absolute Reticulocyte Count <80 x 109/L with Hemoglobin <7.0 gm/dL
   4. Platelets <80 x 109/L
   5. Absolute Neutrophil Count <1.0 x 109/L
5. Found to be with acute illness at enrolment with fever in last 1 week, respiratory infection, etc.
6. History of a sickle crisis within the prior 2 weeks, or blood transfusion within the past 90 days Participants with temporary exclusion can be enrolled later when stable or the excluding criteria has resolved

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 270 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
The frequency, age specific prevalence and severity of Sickle Cell Vasculopathy manifested by New stroke as assessed by the Pediatric NIH Stroke Scale (PedNIHSS) over the 3-year study while on hydroxyurea treatment, compared to baseline assessments. | 3 years
  Baseline assessment will be completed for all study participants and over the 3-year study, scheduled outcome assessments will be performed at study months 18 and 36.
  These assessments will aim to document New (incident) stroke as assessed by the PedNIHSS
The frequency, age specific prevalence and severity of Sickle Cell Vasculopathy manifested by a change in transcranial doppler (TCD) velocity by 15cm/sec or more over the 3-year study while on hydroxyurea treatment, compared to baseline assessment. | 3 years
  Baseline assessment will be completed for all study participants and over the 3-year study, scheduled outcome assessments will be performed at study months 18 and 36.These assessments will aim to document a change in TCD velocity by 15cm/sec or more.
The frequency, age specific prevalence and severity of SCV manifested by New or worsening cognitive impairment, both quantitative and categorical over the 3-year study while on hydroxyurea treatment, compared to baseline assessments. | 3 years
  Baseline assessment will be completed for all study participants and over the 3-year study, scheduled outcome assessments will be performed at study months 18 and 36.These assessments will aim to document new or worsening cognitive impairment - both quantitative and categorical (by standardized criteria ≤-2 z-score) compared to established criteria

SECONDARY OUTCOMES:
Stabilized or worsened structural changes on brain Magnetic Resonance Imaging(MRI) over the 3 years compared to baseline | 3 years
  Brain magnetic resonance will be performed on a subset of subjects at baseline and study month 36 only. Stabilized or worsened structural changes on brain Magnetic Resonance Imaging(MRI) over the 3 years compared to baseline will be assessed.
Stabilized or worsened structural changes on brain Magnetic Resonance Angiography(MRA) over the 3 years compared to baseline | 3 years
  Brain magnetic resonance angiography will be performed on a subset of subjects, at baseline and study month 36 only. Stabilized or worsened structural changes on brain Magnetic Resonance Angiography over the 3 years compared to baseline will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Idro, PhD, Principal Investigator — Makerere University; Nancy Green, MD, Principal Investigator — Columbia University
Locations (1):
- Global Health Uganda, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Provider Investigator- Dr Richard Idro Recipient Investigator- Dr Nancy Green Permitted Uses of Data Set Scientific publication Inform policies Systematic reviews Safety investigations Other legitimate academic and policy issues.
  Data Set Content
  1. Demographic data
  2. Interventional drug data
  3. Cognitive data including all neurocognitive tests administered at 0, 18 and 36 months follow-ups.
  4. Laboratory data including hemograms, haemoglobin electrophoresis, serum chemistry results, inflammatory markers, SCA variants at all scheduled time points.
  5. Neuroimaging data including all MRI data
  6. TCD data
  7. Scheduled visit clinical data including history, physical examination, PedNIHSS at baseline,18 and 36 months.
  8. Unscheduled visits data including all adverse events
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 years

REFERENCES:
- [Background] Galadanci NA, Umar Abdullahi S, Vance LD, Musa Tabari A, Ali S, Belonwu R, Salihu A, Amal Galadanci A, Wudil Jibir B, Bello-Manga H, Neville K, Kirkham FJ, Shyr Y, Phillips S, Covert BV, Kassim AA, Jordan LC, Aliyu MH, DeBaun MR. Feasibility trial for primary stroke prevention in children with sickle cell anemia in Nigeria (SPIN trial). Am J Hematol. 2017 Aug;92(8):780-788. doi: 10.1002/ajh.24770. Epub 2017 Jun 15. PMID 28439953
- [Derived] Naggayi SK, Kalibbala D, Mboizi V, Ssenkusu J, Jin Z, Rosano C, Munube D, Wambaka B, Namazzi R, Kasirye P, Kabatabaazi M, Nambatya G, Murungi S, Nabaggala C, Nakafeero M, Troidl IR, Opoka R, Idro R, Bangirana P, Green NS. Neurocognitive gains among Ugandan children with sickle cell anemia on hydroxyurea: 18-month interim trial results. Blood Adv. 2025 Jun 24;9(12):3116-3127. doi: 10.1182/bloodadvances.2024015073. PMID 40085947
- [Derived] Mboizi V, Nabaggala C, Munube D, Ssenkusu JM, Kasirye P, Kamya S, Kawooya MG, Boehme A, Minja F, Mupere E, Opoka R, Rosano C, Idro R, Green NS. Hydroxyurea therapy for neurological and cognitive protection in pediatric sickle cell anemia in Uganda (BRAIN SAFE II): Protocol for a single-arm open label trial. Contemp Clin Trials Commun. 2024 Nov 28;42:101404. doi: 10.1016/j.conctc.2024.101404. eCollection 2024 Dec. PMID 39717517